CLINICAL TRIAL: NCT05232370
Title: The Effect of Enalapril, Losartan or Not Antihypertensive on the Oxidative Status in Renal Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unidad de Investigacion Medica en Enfermedades Renales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIMER004
Record Dates: First submitted 2022-01-06; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — Angiotensin-Converting Enzyme Inhibitors; Enalapril; Angiotensin Receptor Antagonists; Losartan

STUDY DESIGN:
Intervention Model Description: Three groups are made
  1. - Control group: No treatment
  2. - Tratment group: Enalapril
  3. - Treatment group: Losartan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Recipients of a RT, from a living related donor (DVR) or living unrelated donor (DVNoR) who agreed to participate and signed the Letter of Consent under Information.
  Randomly assigned to control group (Without losartan or enalapril)
- Enalapril group (Experimental): Recipients of a RT, from a living related donor (DVR) or living unrelated donor (DVNoR) who agreed to participate and signed the Letter of Consent under Information.
  Randomly assigned to Enalapril group
  Interventions: Drug: Angiotensin converting enzyme inhibitor
- Losartan group (Experimental): Recipients of a RT, from a living related donor (DVR) or living unrelated donor (DVNoR) who agreed to participate and signed the Letter of Consent under Information.
  Randomly assigned to Losartan group
  Interventions: Drug: Angiotensin Receptor Blockers

INTERVENTIONS:
Drug: Angiotensin converting enzyme inhibitor — Angiotensin-converting enzyme inhibitors after Kidney Transplant
  Other Names: Enalapril
  Arms: Enalapril group
Drug: Angiotensin Receptor Blockers — Angiotensin receptor blockers after Kidney Transplant
  Other Names: Losartan
  Arms: Losartan group

SUMMARY:
The clinical and biochemical improvement observed in kidney transplant (RT) recipients is remarkable. The correct functioning of the allograft depends on various factors such as the donor's age, the alloimmune response, the ischemia-reperfusion injury, arterial hypertension, and the interstitial fibrosis of the allograft, among others. Antihypertensive drugs are necessary for arterial hypertension patients to avoid or reduce the probability of affecting graft function in RT recipients. Oxidative stress (OS) is another complex pathophysiological process with the ability to alter post-transplant kidney function. The study's objective was to determine the effect of the administration of Enalapril, Losartan, or not antihypertensive medication on the oxidative state in RT recipients at the beginning of the study and one year of follow-up.

DETAILED DESCRIPTION:
An open, randomized clinical trial is proposed with a control group. It is carried out in the Transplant Division of the High Specialty Medical Unit of the Hospital de Especialidades, Centro Médico Nacional de Occidente of the Mexican Institute of Social Security in Guadalajara, Jalisco, Mexico. The sample size was based on the formula to evaluate mean differences for clinical trials. Three study groups were formed; thirteen patients with RT who did not require any antihypertensive. Thirteen RT patients to receive Enalapril as an antihypertensive regimen. Thirteen RT patients to receive Losartan as an antihypertensive regimen in the post-transplant period. Recipients of a RT, from a living related donor (DVR) or living unrelated donor (DVNoR) who agreed to participate and signed the Letter of Consent under Information.

Patients who received an RT from a deceased donor, from a donor >55 years, with renal comorbidities at the time of the study (urolithiasis, infections, diabetes), with blood dyscrasias, second transplantation, treatment with non-steroidal anti-inflammatory drugs, statins, spironolactone, pentoxifylline, patients with neurodegenerative processes or who withdrew the Letter of Consent under Information are not eligeble.

ELIGIBILITY:
Inclusion Criteria:

* Renal trasplant, from a living related donor (DVR) or living unrelated donor (DVNoR)
* Who agreed to participate and signed the Letter of Consent under Information.

Exclusion Criteria:

* Patients who received an RT from a deceased donor,
* With donor >55 years,
* With renal comorbidities at the time of the study (urolithiasis, infections, diabetes),
* With blood dyscrasias,
* Second transplantation,
* Those with treatment with non-steroidal anti-inflammatory drugs,
* Treatment with statins, spironolactone, pentoxifylline, patients
* With neurodegenerative processes
* Those who withdrew the Letter of Consent under Information

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
Products of lipoperoxidation (LPO) (oxidative stress molecule) | 1 year after renal transplant
  Measured in mM
Nitric Oxide (NO) (oxidative stress molecule) | 1 year after renal transplant
  Measured in µg/mL

SECONDARY OUTCOMES:
Superoxide dismutase (SOD) (Antioxidative molecule) | 1 year after renal transplant
  Measured in U/L
Glutathione peroxidase (GPx) (Antioxidative molecule) | 1 year after renal transplant
  Measured in nmol/min/mL
Total Antioxidant Capacity (TAC) (Antioxidative molecule) | 1 year after renal transplant
  Measured in µM

CONTACTS AND LOCATIONS:
Locations (1):
- Enrique Rojas Campos, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No